CLINICAL TRIAL: NCT04490915
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Crinecerfont (NBI-74788) in Adult Subjects With Classic Congenital Adrenal Hyperplasia, Followed by Open-Label Treatment
Brief Title: Global Safety and Efficacy Registration Study of Crinecerfont for Congenital Adrenal Hyperplasia
Acronym: CAHtalyst
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-74788-CAH3003; 2019-004873-17 (EudraCT Number); 2023-509171-16-00 (EU CTIS Number)
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — crinecerfont

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule, administered orally, twice daily for 24 weeks, followed by active treatment with crinecerfont for at least 1 year.
  Interventions: Drug: Crinecerfont; Drug: Placebo
- Crinecerfont (Experimental): Crinecerfont capsule, administered orally, twice daily for 24 weeks during the placebo-controlled treatment period, followed by active treatment with crinecerfont for at least 1 year.
  Interventions: Drug: Crinecerfont

INTERVENTIONS:
Drug: Crinecerfont — CRF type 1 receptor antagonist
  Other Names: NBI-74788; Crenessity
Drug: Placebo — Non-active dosage form
  Arms: Placebo

SUMMARY:
This is a Phase 3 study to evaluate the efficacy, safety, and tolerability of crinecerfont versus placebo administered for 24 weeks in approximately 165 adult participants with classic CAH due to 21-hydroxylase deficiency. The study consists of a 24-week randomized, double-blind, placebo-controlled period, followed by 1 year of active treatment with crinecerfont. Subsequently, participants may elect to participate in the open-label extension (OLE) period. The duration of participation in the study is approximately 20 months for the core study and will be a variable amount of time per participant for the OLE (estimated to be approximately 3 years).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to adhere to the study procedures, including all requirements at the study center and return for the follow-up visit.
2. Have a medically confirmed diagnosis of classic CAH due to 21-hydroxylase deficiency.
3. Be on a stable steroid regimen.
4. Participants of childbearing potential must agree to use an acceptable method of contraception during the study.

Exclusion Criteria:

1. Have a diagnosis of any of the other known forms of classic CAH.
2. Have a history of bilateral adrenalectomy, hypopituitarism, or other condition requiring chronic glucocorticoid therapy.
3. Have a clinically significant unstable medical condition or chronic disease other than CAH.
4. Have a history of cancer unless considered cured.
5. Are pregnant.
6. Have a known history of clinically significant arrhythmia or abnormalities on ECG.
7. Have a known hypersensitivity to any corticotropin releasing hormone receptor antagonists.
8. Have received any other investigational drug within 30 days before initial screening or plan to use an investigational drug (other than the study drug) during the study.
9. Have current substance dependence, or current substance (drug) or alcohol abuse.
10. Have had a blood loss ≥550 mL or donated blood or blood products within 8 weeks prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2027-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (65):
- United States (20):
  - Neurocrine Clinical Site, Los Angeles, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, San Francisco, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Indianapolis, Indiana
  - Neurocrine Clinical Site, Bethesda, Maryland
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Minneapolis, Minnesota
  - Neurocrine Clinical Site, Rochester, Minnesota
  - Neurocrine Clinical Site, St Louis, Missouri
  - Neurocrine Clinical Site, Great Neck, New York
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, Winston-Salem, North Carolina
  - Neurocrine Clinical Site, Tulsa, Oklahoma
  - Neurocrine Clinical Site, Philadelphia, Pennsylvania
  - Neurocrine Clinical Site, Pittsburgh, Pennsylvania
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Seattle, Washington
- Austria (2):
  - Neurocrine Clinical Site, Graz
  - Neurocrine Clinical Site, Vienna
- Belgium (2):
  - Neurocrine Clinical Site, Brussels
  - Neurocrine Clinical Site, Leuven
- Neurocrine Clinical Site, Sofia, Bulgaria
- Neurocrine Clinical Site, Halifax, Nova Scotia, Canada
- Neurocrine Clinical Site, Hradec Králové, Czechia
- France (5):
  - Neurocrine Clinical Site, Angers
  - Neurocrine Clinical Site, Grenoble
  - Neurocrine Clinical Site, Le Kremlin-Bicêtre
  - Neurocrine Clinical Site, Nantes
  - Neurocrine Clinical Site, Paris
- Germany (5):
  - Neurocrine Clinical Site, Dresden
  - Neurocrine Clinical Site, Essen
  - Neurocrine Clinical Site, Frankfurt
  - Neurocrine Clinical Site, Leipzig
  - Neurocrine Clinical Site, Munich
- Greece (2):
  - Neurocrine Clinical Site, Athens
  - Neurocrine Clinical Site, Thessaloniki
- Israel (4):
  - Neurocrine Clinical Site, Afula
  - Neurocrine Clinical Site, Beersheba
  - Neurocrine Clinical Site, Petah Tikva
  - Neurocrine Clinical Site, Tel Aviv
- Italy (8):
  - Neurocrine Clinical Site, Ancona
  - Neurocrine Clinical Site, Bologna
  - Neurocrine Clinical Site, Florence
  - Neurocrine Clinical Site, Messina
  - Neurocrine Clinical Site, Milan
  - Neurocrine Clinical Site, Naples
  - Neurocrine Clinical Site, Padua
  - Neurocrine Clinical Site, Roma
- Neurocrine Clinical Site, Leiden, Netherlands
- Poland (3):
  - Neurocrine Clinical Site, Krakow
  - Neurocrine Clinical Site, Poznan
  - Neurocrine Clinical Site, Warsaw
- Neurocrine Clinical Site, Porto, Portugal
- Neurocrine Clinical Site, Belgrade, Serbia
- Spain (2):
  - Neurocrine Clinical Site, Madrid
  - Neurocrine Clinical Site, Seville
- Sweden (2):
  - Neurocrine Clinical Site, Gothenburg
  - Neurocrine Clinical Site, Stockholm
- United Kingdom (4):
  - Neurocrine Clinical Site, Cardiff
  - Neurocrine Clinical Site, London
  - Neurocrine Clinical Site, Manchester
  - Neurocrine Clinical Site, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Auchus RJ, Hamidi O, Pivonello R, Bancos I, Russo G, Witchel SF, Isidori AM, Rodien P, Srirangalingam U, Kiefer FW, Falhammar H, Merke DP, Reisch N, Sarafoglou K, Cutler GB Jr, Sturgeon J, Roberts E, Lin VH, Chan JL, Farber RH; CAHtalyst Adult Trial Investigators. Phase 3 Trial of Crinecerfont in Adult Congenital Adrenal Hyperplasia. N Engl J Med. 2024 Aug 8;391(6):504-514. doi: 10.1056/NEJMoa2404656. Epub 2024 Jun 1. PMID 38828955
- See also: Study website - CAHtalyst Study — https://www.cahtalyststudy.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study includes a double-blind (DB) placebo-controlled treatment period, an open-label (OL) treatment period, an OL or DB active-controlled treatment period, and an open-label extension (OLE) treatment period. The study is ongoing. Only the primary analysis results (as of 19 July 2023 data cutoff date) have been reported. The final results will be reported after completion of the study.
Groups:
- Placebo: Participants received crinecerfont-matched placebo orally twice daily for 24 weeks during the DB placebo-controlled treatment period. After the 24-week DB placebo-controlled treatment period, there was a 6-month, OL treatment period, during which all participants received crinecerfont.
- Crinecerfont: Participants received crinecerfont orally twice daily for 24 weeks during the DB placebo-controlled treatment period. After the 24-week DB placebo-controlled treatment period, there was a 6-month, OL treatment period, during which all participants received crinecerfont.
Period: DB Treatment Period (24 Weeks)
Arm/Group | Placebo | Crinecerfont
Started | 60 | 122
Received at Least 1 Dose of Study Drug | 59 | 122
Completed | 57 | 117
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 0 | 1
Period: OL Treatment Period (6 Months)
Arm/Group | Placebo | Crinecerfont
Started | 57 | 117
Received at Least 1 Dose of Study Drug | 57 | 117
Completed | 22 | 57
Not Completed | 35 | 60
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Ongoing in the Study | 34 | 58

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Crinecerfont | Total
Number analyzed (Participants) | 60 | 122 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (10.17) | 31.3 (9.82) | 30.8 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 61 | 90
  Male | 31 | 61 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 52 | 116 | 168
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 57 | 107 | 164
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 6 | 8
Daily Glucocorticoid Dose [Mean (Standard Deviation); unit: milligrams (mg)/day] | 32.06 (32.06) | 32.44 (9.24) | 32.31 (9.30)
Daily Glucocorticoid Dose Adjusted for Body Surface Area [Mean (Standard Deviation); unit: mg/square meter (m^2)/day] | 17.91 (5.45) | 17.45 (4.54) | 17.60 (4.85)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Glucocorticoid Daily Dose at Week 24
Description: Least square (LS) mean and standard error (SE) were calculated using analysis of covariance (ANCOVA) model.
Time Frame: Baseline, Week 24
Population: Full Analysis Set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo: Participants received crinecerfont-matched placebo orally twice daily for 24 weeks during the DB placebo-controlled treatment period.
- Crinecerfont: Participants received crinecerfont orally twice daily for 24 weeks during the DB placebo-controlled treatment period.
Arm/Group | Placebo | Crinecerfont
Number analyzed (Participants) | 60 | 122
percent change | -10.300 (3.247) | -27.322 (2.418)
Statistical Analysis 1: Comparison: Placebo vs Crinecerfont; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -17.022, 95% CI 2-sided [-23.802 to -10.243], Standard Error of Mean 3.433 — LS Mean Difference of Crinecerfont - Placebo

2. Secondary Outcome: Change From Baseline in Serum Androstenedione at Week 4
Time Frame: Baseline, Week 4
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants Who Achieved a Reduction to Physiologic Glucocorticoid Dose While Maintaining Androstenedione Control at Week 24
Time Frame: Week 24
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

5. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Percent Total Fat Mass at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in Serum 17-hydroxyprogesterone (17-OHP) at Week 4
Time Frame: Baseline, Week 4
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in Blood Pressure at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in Glucose Tolerance at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in Waist Circumference at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline in Menstrual Regularity at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline in Testicular Adrenal Rest Tumor (TART) Volume at Week 24
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: Per planned analysis all-cause mortality data were collected and reported for all randomized participants. Adverse events (serious and other) were collected and reported for all randomized participants who received at least 1 dose of study drug. Only DB period was complete at the time of data cutoff date.
Groups:
- DB Period: Placebo: Participants received crinecerfont-matched placebo orally twice daily for 24 weeks during the DB placebo-controlled treatment period.
- DB Period: Crinecerfont: Participants received crinecerfont orally twice daily for 24 weeks during the DB placebo-controlled treatment period.
Arm/Group | DB Period: Placebo | DB Period: Crinecerfont
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/59 | 4/122
Other Adverse Events (participants affected / at risk) | 39/59 | 76/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=59) | DB Period: Crinecerfont (N=122)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=59) | DB Period: Crinecerfont (N=122)
Fatigue (General disorders) | 9 | 30
Headache (Nervous system disorders) | 9 | 19
Coronavirus infection (Infections and infestations) | 5 | 17
Upper respiratory tract infection (Infections and infestations) | 7 | 11
Diarrhoea (Gastrointestinal disorders) | 5 | 10
Dizziness (Nervous system disorders) | 2 | 10
Nausea (Gastrointestinal disorders) | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Pyrexia (General disorders) | 6 | 7
Nasopharyngitis (Infections and infestations) | 8 | 6
Vomiting (Gastrointestinal disorders) | 5 | 6
Anxiety (Psychiatric disorders) | 5 | 4
Acne (Skin and subcutaneous tissue disorders) | 4 | 4
Urinary tract infection (Infections and infestations) | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Asthenia (General disorders) | 5 | 2
Blood androstenedione increased (Investigations) | 3 | 2
Renin increased (Investigations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04490915/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT04490915/SAP_001.pdf